CLINICAL TRIAL: NCT05790434
Title: Investigation on Diagnostic Criteria for Septic Arthritis：a Multi-center Nested Case-control Study
Brief Title: Diagnostic Criteria for Septic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0909
Record Dates: First submitted 2023-02-07; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Septic Arthritis
Keywords: Septic Arthritis; diagnostic criteria
MeSH Terms: conditions — Arthritis, Infectious | interventions — Clinical Laboratory Techniques; Physical Examination; Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with septic arthritis
  Interventions: Diagnostic Test: Laboratory test; Diagnostic Test: History taking and physical examination; Diagnostic Test: biopsy
- Controls: Patients with osteoarthritis, rheumatoid arthritis
  Interventions: Diagnostic Test: Laboratory test; Diagnostic Test: History taking and physical examination; Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: Laboratory test — including white blood cell count, C-reactive protein, erythrocyte sedimentation rate, percent of polymorphonuclear leukocytes, albumin, and globulin
Diagnostic Test: History taking and physical examination — including fever, joint pain, local swelling and redness, sinus
Diagnostic Test: biopsy — including arthrocentesis culture，and frozen section

SUMMARY:
Septic arthritis (SA) is a rare but highly disabling disease. The ideal diagnosis criteria is not well established. There is an urgent need to establish golden standard for diagnosis.

DETAILED DESCRIPTION:
Septic arthritis (SA) is a rare but highly disabling disease. Epidemiologic studies have documented an incidence of 0.9-1.3 per 100,000 [1, 2]. The treatment is challenging and the ideal diagnosis criteria is not well established. The specific tactics employed by relevant researches varied widely [3-6]. Patients with recurrent sepsis may require arthrodesis or amputation, which would result in severe functional loss [2]. Therefore, there is an urgent need to establish golden standard for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* admission to orthopaedics
* complete data

Exclusion Criteria:

* Accompanied with fracture
* Accompanied with other infections
* Accompanied with immune system diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: general hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
WBC counts | preoperatively
  white blood cell (WBC) counts
%PMN | preoperatively
  percent of polymorphonuclear leukocytes (%PMN)
CRP | preoperatively
  concentration of C-reactive protein (CRP)
ESR | preoperatively
  erythrocyte sedimentation rate (ESR)
Albumin | preoperatively
  concentration of albumin
Globulin | preoperatively
  concentration of globulin
Body temperature | preoperatively
  to check whether there has been a fever (>37.2°C) previously or now by medical history consultation and physical examination
joint swelling and redness | preoperatively
  to check whether there is joint swelling and redness by visual inspection and palpation
sinus tract | preoperatively
  to check whether there is any sinus tract by visual inspection
positive X-ray findings | preoperatively
  to determine whether there are positive X-ray findings, such as bone destruction, narrowing of the joint space, etc.
positive MR findings | preoperatively
  to determine whether there are positive MR findings, such as joint effusion, cartilage damage, etc.
positive pathological findings | intraoperatively
  determined by 5 or more neutrophils per high-power field on histopathologic examination
positive culture | preoperatively
  determined by a bacterial growth when culture of blood or joint fluid in agarose

CONTACTS AND LOCATIONS:
Overall Officials: Lan Tang, MD, Study Director — School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - Zhejiang hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross JJ. Septic Arthritis of Native Joints. Infect Dis Clin North Am. 2017 Jun;31(2):203-218. doi: 10.1016/j.idc.2017.01.001. Epub 2017 Mar 30. PMID 28366221
- [Background] Abram SGF, Alvand A, Judge A, Beard DJ, Price AJ. Mortality and adverse joint outcomes following septic arthritis of the native knee: a longitudinal cohort study of patients receiving arthroscopic washout. Lancet Infect Dis. 2020 Mar;20(3):341-349. doi: 10.1016/S1473-3099(19)30419-0. Epub 2019 Dec 17. PMID 31862240
- [Background] Mathews CJ, Weston VC, Jones A, Field M, Coakley G. Bacterial septic arthritis in adults. Lancet. 2010 Mar 6;375(9717):846-55. doi: 10.1016/S0140-6736(09)61595-6. PMID 20206778
- [Background] Padaki AS, Ma GC, Truong NM, Cogan CJ, Lansdown DA, Feeley BT, Ma CB, Zhang AL. Arthroscopic Treatment Yields Lower Reoperation Rates than Open Treatment for Native Knee but Not Native Shoulder Septic Arthritis. Arthrosc Sports Med Rehabil. 2022 May 27;4(3):e1167-e1178. doi: 10.1016/j.asmr.2022.04.014. eCollection 2022 Jun. PMID 35747656
- [Background] Johns BP, Loewenthal MR, Dewar DC. Open Compared with Arthroscopic Treatment of Acute Septic Arthritis of the Native Knee. J Bone Joint Surg Am. 2017 Mar 15;99(6):499-505. doi: 10.2106/JBJS.16.00110. PMID 28291183
- [Background] Shaikh AA, Ha CW, Park YG, Park YB. Two-stage approach to primary TKA in infected arthritic knees using intraoperatively molded articulating cement spacers. Clin Orthop Relat Res. 2014 Jul;472(7):2201-7. doi: 10.1007/s11999-014-3545-6. Epub 2014 Mar 6. PMID 24599649